CLINICAL TRIAL: NCT05745883
Title: A Phase 1b Multicenter, Randomized, Double-Blind, Placebo-Controlled Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DISC-0974 in Participants With Non-Dialysis Dependent Chronic Kidney Disease and Anemia
Brief Title: Study of DISC-0974 to Assess the Safety, Tolerability, PK and PD of DISC-0974 in Participants With CKD and Anemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Disc Medicine, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DISC-0974-103
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; Anemia of Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b Single Dose (Experimental): Single dose of DISC-0974
- Single Dose of Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo
- Phase 1b Multiple Doses (Experimental): Multiple doses of DISC-0974
  Interventions: Drug: DISC-0974
- Multiple Doses of Placebo (Placebo Comparator): Multiple doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DISC-0974 — DISC-0974 is administered subcutaneously
  Arms: Phase 1b Multiple Doses
Drug: Placebo — Placebo is administered subcutaneously
  Arms: Multiple Doses of Placebo; Single Dose of Placebo

SUMMARY:
This Phase 1b study of DISC-0974 will assess the safety, tolerability, pharmacokinetics (PK) and Pharmacodynamics (PD) of DISC-0974 in adult participants with Non-Dialysis Dependent Chronic Kidney Disease and Anemia.

ELIGIBILITY:
Inclusion criteria:

1. Aged ≥18 years of age at the time of signing informed consent.
2. Non-dialysis-dependent chronic kidney disease, Stages 2-5, defined as eGFR <90 mL/min/1.73 m2 using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
3. Hgb <11.0 g/dL
4. Serum ferritin ≥50 μg/L at screening
5. Transferrin saturation ≤35%
6. AST and ALT <2× upper limit of normal (ULN) at screening
7. Total and direct bilirubin <ULN at screening
8. If female, then EITHER postmenopausal, defined as at least 12 months of natural, spontaneous amenorrhea and serum follicle-stimulating hormone >40 mIU/mL at screening, or at least 6 weeks following surgical menopause (bilateral oophorectomy or hysterectomy); OR agreeable to use of highly effective contraception (listed below) on Day 1 (or earlier) for at least 8 weeks after the last dose of study drug:

   * Stable hormonal contraceptive (≥3 months) in conjunction with a barrier method (eg, condom [male or female] or diaphragm)
   * Intrauterine device in place for at least 3 months
   * Tubal ligation or single male partner with vasectomy in conjunction with a barrier method (eg, condom [male or female] or diaphragm)
9. If male with female sexual partner(s) of childbearing potential, agrees to use one of the following acceptable methods of contraception during the study and for at least 8 weeks after the last study drug dose:

   1. Stable hormonal contraceptive (≥3 months; female partner) in conjunction with a barrier method (eg, condom or diaphragm [female partner])
   2. Intrauterine device in place for at least 3 months (female partner)
   3. Surgically sterile hysterectomy, bilateral oophorectomy, or bilateral tubal ligation (female partner) in conjunction with a barrier method (eg, condom [male or female] or diaphragm)
   4. Confirmed successful vasectomy in conjunction with a barrier method (eg, condom [male or female] or diaphragm)
10. Able to understand and provide written informed consent
11. Able to comply with all study procedures

Exclusion Criteria:

1. Treatment within 2 days prior to screening with oral iron or iron-containing supplements. Participants may be considered for the study if they undergo a 2-day washout period prior to signing the informed consent form (ICF) and screening for oral iron or iron-containing supplements. Between screening and 2 days prior to baseline visit, participants may continue oral iron or iron-containing supplements at the discretion of the Investigator, but any study-related lab draws will require a 48-hour washout from oral iron
2. Treatment within 30 days prior to screening with one of the following anemia treatments: blood transfusion, ESAs, or IV iron. Participants may be considered for the study if they undergo a 30-day washout period prior to signing the ICF and screening for erythropoietin-stimulating agents or IV iron
3. Acute dialysis or acute kidney injury within 12 weeks prior to screening or expected need to start dialysis within 24 weeks of screening
4. Hospitalization for a CV, renal, or cardiorenal condition within 30 days prior to screening
5. Positive direct antiglobulin test with reactive eluate at screening or active hemolytic anemia. This test can be performed prior to other screening procedures after the participant is consented for the prescreening testing
6. History of hereditary hemochromatosis
7. History of hemoglobinopathy or intrinsic red blood cell defect associated with anemia
8. History of total splenectomy
9. Hematopoietic stem cell or solid organ transplant within the past 10 years
10. Medical history of anemia from B12 or folate deficiency, infection, or bleeding in the 3 months prior to screening
11. Stroke, myocardial infarction, deep venous thrombosis, pulmonary or arterial embolism within 6 months prior to screening
12. If female, pregnant or breastfeeding
13. Any major surgery within 8 weeks before screening or incomplete recovery from any previous surgery
14. History of malignancy within the last 3 years. The following history/concurrent conditions are allowed: basal or squamous cell carcinoma skin cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast, histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system). A history of completed treatment (medical or surgical) of Stage 1-2 cancers may be permitted with prior Sponsor agreement
15. Participation in any other clinical protocol or investigational study that involves administration of experimental therapy and/or therapeutic devices within 30 days of screening
16. A history or known allergic reaction to any investigational product excipients or history of anaphylaxis to any food or drug
17. History of anti-drug antibody formation
18. History of inadequately controlled heart disease (New York Heart Association Classification 3 or 4) and/or have a known left ventricular ejection fraction <35%
19. Uncontrolled fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement, despite appropriate treatment)
20. Human immunodeficiency virus positive, active hepatitis B, or active hepatitis C
21. Uncontrolled diabetes mellitus (defined as diabetes mellitus requiring initiation of insulin therapy within 3 months of screening)
22. Significant medical condition, laboratory abnormality, or psychiatric condition that would prevent the patient from participating in the study
23. Any condition or concomitant medication that would confound the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | up to 145 days
Incidence of clinically abnormal vital signs | up to 145 days
Incidence of abnormal laboratory test results | up to 145 days
Incidence of clinically abnormal physical exam | up to 145 days
Incidence of clinically abnormal electrocardiograms | up to 145 days

SECONDARY OUTCOMES:
Change from baseline in concentration of iron laboratory parameter | up to 145 days
Change from baseline in concentration of hematologic laboratory parameters | up to 145 days
Cmax-Maximum drug concentration measured in plasma | up to 145 days
Tmax-Time of maximum drug concentration | up to 145 days
AUC-Area under the drug concentration time curve | up to 145 days
T½ - Elimination half life of the drug | up to 145 days
CL/F-Apparent drug clearance (only for single-dose portion) | up to 57 days
Vz/F; Vss/F -Apparent volume of distribution of the drug (only for single-dose portion) | up to 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Will Savage, MD PhD, Study Director — Disc Medicine
Locations (13):
- United States (13):
  - UCLA Clinical and Translational Research, Los Angeles, California
  - US Renal Care Inc., Lone Tree, Colorado
  - Accel Research, DeLand, Florida
  - Total Research Group, Miami, Florida
  - Flourish Research, Winter Park, Florida
  - Nephrology and Hypertension Specialists, PC-Dalton, Dalton, Georgia
  - CARE Institute - Boise Kidney, Boise, Idaho
  - Center for Advanced Kidney Research PLC, Saint Clair Shores, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Centricity Research, Columbus, Ohio
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Washington Nephrology Associates, LLP, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: No